CLINICAL TRIAL: NCT06272838
Title: The Effectiveness of the Exercise Program Applied With the Biodex Balance System in Patients With Parkinson's Disease
Brief Title: Biodex Balance System in Patients With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, Principal Investigator, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-19/145
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Balance training; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Randomised controlled
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes Assessor will be different persons
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In addition to conventional balance exercises, the exercise program, which includes games to improve balance, performed with the help of a Biodex balance device, will be given in a total of 20 sessions, 5 days a week, for 4 weeks..
  Interventions: Other: Biodex balance system; Other: The conventional balance exercise program
- Control Group (Active Comparator): The conventional balance exercise program will be applied by a physiotherapist for 4 weeks, 5 days a week, in a total of 20 sessions.
  Interventions: Other: The conventional balance exercise program

INTERVENTIONS:
Other: Biodex balance system — In addition to the conventional exercise program, it will be applied on a platform with the Biodex balance system for 4 weeks, 5 days a week, in a total of 20 sessions.
  Arms: Experimental Group
Other: The conventional balance exercise program — The conventional balance exercise program will be applied by a physiotherapist for 4 weeks, 5 days a week, in a total of 20 sessions.

SUMMARY:
Conventional balance exercises are an effective rehabilitation method applied in routine rehabilitation programs for Parkinson's patients. With technological developments, balance exercises

DETAILED DESCRIPTION:
This study was planned based on the hypothesis that exercises based on visual feedback applied to patients through games will increase patient compliance and improve balance better than conventional exercise.Previous studies have shown that the Biodex balance device has positive contributions to balance in neurological and orthopedic rehabilitation applications.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's diagnosis and Hoehn Yahr stage I-III
* Not changing medical treatment in the last three months
* Mini mental test score is over twenty-four

Exclusion Criteria:

* Vestibular hypofunction
* Neurological disease other than Parkinson's disease (multiple sclerosis, stroke, myopathy)
* History of lower extremity surgery (such as arthroplasty, anterior cruciate ligament repair)
* Upper limb amputation in the participant
* Impairment in cognitive functions
* History of psychotic illness
* Presence of stage 4 gonarthrosis history of malignancy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-28 (Estimated); Primary Completion 2024-09-14 (Estimated); Study Completion 2024-10-14 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline
  Berg Balance Scale was developed to measure balance performance and is used to evaluate postural control and predict fall risk. Higher scores indicate better balance
Berg Balance Scale | 4th week
  Berg Balance Scale was developed to measure balance performance and is used to evaluate postural control and predict fall risk. Higher scores indicate better balance
Berg Balance Scale | 8 th week
  Berg Balance Scale was developed to measure balance performance and is used to evaluate postural control and predict fall risk. Higher scores indicate better balance
Biodex dynamic balance score | Baseline
  The balance assessment of the participants will be made with the Biodex Balance Systems device. During the measurement, patients will try to stay balanced on the device whose platform stability is adjusted.
Biodex dynamic balance score | 4th week
  The balance assessment of the participants will be made with the Biodex Balance Systems device. During the measurement, patients will try to stay balanced on the device whose platform stability is adjusted.
Biodex dynamic balance score | 8th week
  The balance assessment of the participants will be made with the Biodex Balance Systems device. During the measurement, patients will try to stay balanced on the device whose platform stability is adjusted.
The fall efficacy scale | Baseline
  The fall efficacy scale consists of 10 questions rated on a 10-point Likert scale. Getting more than 70 points from the scale indicates fear of falling.
The fall efficacy scale | 4th week
  The fall efficacy scale consists of 10 questions rated on a 10-point Likert scale. Getting more than 70 points from the scale indicates fear of falling.
The fall efficacy scale | 8th week
  The fall efficacy scale consists of 10 questions rated on a 10-point Likert scale. Getting more than 70 points from the scale indicates fear of falling.
Time up and go test | Baseline
  Time up and go testing will be performed to determine fall risk and measure balance, sit-to-stand and walking progress. Minimal detectable change in Parkinson's patients. It is 3.5 seconds. (10.2522/ptj.20090126.)
Time up and go test | 4th week
  Time up and go testing will be performed to determine fall risk and measure balance, sit-to-stand and walking progress. Minimal detectable change in Parkinson's patients. It is 3.5 seconds. (10.2522/ptj.20090126.)
Time up and go test | 8th week
  Time up and go testing will be performed to determine fall risk and measure balance, sit-to-stand and walking progress. Minimal detectable change in Parkinson's patients. It is 3.5 seconds. (10.2522/ptj.20090126.)

SECONDARY OUTCOMES:
The 8-item version of the Parkinson's Disease Questionnaire (PDQ-8) | Baseline
  The 8-item version of the Parkinson's Disease Questionnaire (PDQ-8)is a shortened version of the 39-item Parkinson's Disease Questionnaire (PDQ-39). It is a patient-reported outcome measure used to measure people's quality of life. It consists of 8 questions, each question is scored between 0-4. Higher scores indicate worse quality of life.
The 8-item version of the Parkinson's Disease Questionnaire (PDQ-8) | 4th week
  The 8-item version of the Parkinson's Disease Questionnaire (PDQ-8)is a shortened version of the 39-item Parkinson's Disease Questionnaire (PDQ-39). It is a patient-reported outcome measure used to measure people's quality of life. It consists of 8 questions, each question is scored between 0-4. Higher scores indicate worse quality of life.
The 8-item version of the Parkinson's Disease Questionnaire (PDQ-8) | 8th week
  The 8-item version of the Parkinson's Disease Questionnaire (PDQ-8)is a shortened version of the 39-item Parkinson's Disease Questionnaire (PDQ-39). It is a patient-reported outcome measure used to measure people's quality of life. It consists of 8 questions, each question is scored between 0-4. Higher scores indicate worse quality of life.
The Five Times Sit to Stand Test | 8th week
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements. The patient is asked to stand up quickly and sit down 5 times and the time is recorded.
The Five Times Sit to Stand Test | 4th week
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements. The patient is asked to stand up quickly and sit down 5 times and the time is recorded.
The Five Times Sit to Stand Test | baseline
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements. The patient is asked to stand up quickly and sit down 5 times and the time is recorded.
Beck Depression Inventory | baseline
  Beck depression inventory can be self-scored. It consists of 21 questions. Higher scores indicate increased depression.
Beck Depression Inventory | 4th week
  Beck depression inventory can be self-scored. It consists of 21 questions. Higher scores indicate increased depression.
Beck Depression Inventory | 8th week
  Beck depression inventory can be self-scored. It consists of 21 questions. Higher scores indicate increased depression.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Asst Prof, Principal Investigator — Kirsehir Ahi Evran University
Locations (1):
- Kırşehir Ahi Evran University Faculty of Medicine, Kırşehir, City Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramos GS, Silva-Batista C, Palma BP, Ugrinowitsch C, Cunha TFD. Risk of falls using the Biodex Balance System in non-faller patients with Parkinson Disease. Somatosens Mot Res. 2022 Jun-Dec;39(2-4):111-115. doi: 10.1080/08990220.2021.2018295. Epub 2021 Dec 21. PMID 34930080
- [Background] de Oliveira Lira JL, Ugrinowitsch C, Fecchio R, Coelho DB, Moreira-Neto A, Germano R, de Lima Miliatto AC, Dos Santos Vieira Yano BC, Silva-Batista C. Minimal Detectable Change for Balance Using the Biodex Balance System in Patients with Parkinson Disease. PM R. 2020 Mar;12(3):281-287. doi: 10.1002/pmrj.12216. Epub 2019 Aug 23. PMID 31278834